CLINICAL TRIAL: NCT06652438
Title: Randomized Study to Assess Revumenib in Combination With Azacitidine + Venetoclax in Adult Patients With Newly Diagnosed NPM1-mutated or KMT2A-rearranged AML Ineligible for Intensive Chemotherapy
Brief Title: Revumenib in Combination With Azacitidine + Venetoclax in Patients NPM1-mutated or KMT2A-rearranged AML
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Collaborators: German-Austrian Acute Myeloid Leukemia Study Group (Unknown); United Kingdom AML Research Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HO177; 2024-512733-32-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-02; First posted 2024-10-22 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Acute Myeloid Leukemia, Adult
Keywords: newly AML diagnosed; NPM1; KMT2A
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — revumenib

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Revumenib-placebo (Placebo Comparator): day 1-28 Placebo
  Treatment will be on a continuous 28-day cycle schedule and continued until disease progression, development of unacceptable toxicity, death, withdrawal by subject or other protocol defined criteria for discontinuation (whichever comes first).
  Interventions: Drug: Placebo
- Revumenib (Experimental): day 1-28 Revumenib
  Treatment will be on a continuous 28-day cycle schedule and continued until disease progression, development of unacceptable toxicity, death, withdrawal by subject or other protocol defined criteria for discontinuation (whichever comes first).
  Interventions: Drug: Revumenib

INTERVENTIONS:
Drug: Revumenib — day 1- 28 per cycle
  Arms: Revumenib
Drug: Placebo — day 1- 28 per cycle
  Arms: Revumenib-placebo

SUMMARY:
Treatment of patients with newly diagnosed AML who are not eligible for intensive chemotherapy has remained an area of high unmet medical need. The combination therapy with two medicines, azacitidine and venetoclax, is the usual plan of action. This has brought significant progress in the treatment, but it nevertheless is not curative and the disease does relapse over time.

Revumenib blocks a specific molecule called menin in the cell nucleus. Some types of AML are reliant on menin working properly. These are leukemia cells with a change in the DNA, i.e. a mutation in the NPM1 or KMT2A gene. Revumenib can prevent the production of these types of leukemia cells by disrupting the production of this menin.

The current study investigates whether adding revumenib to the combination therapy improves the prognosis for AML patients with a mutation in the NPM1 or KMT2A gene.

This is a randomized, double-blind, placebo-controlled clinical study where subjects will be treated until disease progression, or development of side effects or death. From the moment of inclusion of the last patient, there will be a 4-year observational follow-up study in order to register survival duration and follow-up visits.

Approximately 415 previously untreated patients with a mutation in the NPM1 or KMT2A gene and with newly diagnosed AML, who are not eligible for intensive chemotherapy. Patients must be ≥18 years of age.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a patient must meet all of the following criteria:

1. Patient with newly diagnosed NPM1-mutated AML, consistent with NPM1c, according to the 2022 International Consensus Classification (i.e. ≥ 10% blasts).

   OR Patient with newly diagnosed KMT2A-rearranged AML according to the 2022 International Consensus Classification (i.e. ≥ 10% blasts). KMT2A partial tandem duplications or deletions are NOT eligible.

   Of note: in case both NPM1 and IDH1 are mutated and both EVOLVE-1 (HO173) and EVOLVE-2 (HO177) are open for inclusion at your site, then patients can only be included in the EVOLVE-1 trial (HO173)
2. Central confirmation of NPM1 mutation or KMT2A rearrangement in one of the dedicated central genetic laboratories.
3. Age ≥ 18 years, no upper age limit.
4. Patient is ineligible for intensive induction chemotherapy by meeting at least 1 of the following criteria:

   * ≥ 75 years of age: ineligible for intensive chemotherapy per physician's discretion (with an ECOG performance status 0-2) .
   * 18-74 years: patient is not eligible for standard chemotherapy because any of the following co-morbidities: o ECOG performance status 2 or 3 .

     * Cardiac history of chronic heart failure requiring treatment; or with an ejection fraction ≤50%; or chronic stable angina.
     * DLCO ≤ 65% or FEV1 ≤ 65%.
     * Creatinine clearance ≥ 30 mL/min to <45 ml/min calculated by the Cockcroft Gault formula.
     * Moderate hepatic impairment with total bilirubin > 1.5 to < 3.0 x upper limit of normal (ULN).
     * Any other comorbidity that the local physician assesses to be incompatible with intensive chemotherapy must be reviewed and approved by the Sponsor's (co-) Principal Investigator (written approval must be sent to HO177@erasmusmc.nl before study enrolment).
5. Patient must have a projected life expectancy of at least 12 weeks (as assessed by the treating physician).
6. Patient must have a white cell blood (WBC) count of < 25 x 109/L. Hydroxyurea can be used prior to study enrolment to reduce the WBC count to meet this criterion.
7. Adequate renal function as evidenced by serum creatinine ≤ 2.0 × upper limit of norm (ULN) or creatinine clearance >30 mL/min based on the Cockcroft-Gault glomerular filtration rate (GFR).
8. Adequate hepatic function as evidenced by:

   * Serum total bilirubin ≤ 3.0 × ULN unless considered due to Gilbert's disease, or leukemic involvement following written approval by the sponsor (Co-)Principal Investigator (copy in HO177@erasmusmc.nl).
   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 3.0 × ULN, unless considered due to leukemic involvement following written approval by the sponsor (Co-)Principal Investigator (copy in HO177@erasmusmc.nl).
9. Female patient must:

   * be of nonchildbearing potential:

     o postmenopausal (defined as at least 1 year without any menses).

     o documented surgically sterile (e.g. documented hysterectomy, bilateral oophorectomy, bilateral salpingectomy or congenital sterile) or status post hysterectomy (at least 1 month prior to screening).
   * or, if of childbearing potential (not surgically sterile and not postmenopausal) agree to avoid pregnancy during the study and for 6 months after the final study drug administration.

     o and have a negative urine or serum pregnancy test at screening.

     o and, if heterosexually active, agree to consistently apply one highly effective* method of birth control in combination to a barrier method for the duration of the study and for 6 months after the final study drug administration.

     *Highly effective forms of birth control include

     - Consistent and correct usage of established hormonal contraceptives that inhibit ovulation for at least 1 month prior to taking study drug. (hormonal contraception is only a highly effective method of birth control, if a combined [estrogen and progestogen containing] hormonal contraception or a progestogen-only hormonal contraception - both associated with inhibition of ovulation - is used.

     - Established intrauterine device (IUD) or intrauterine system (IUS)

     - Bilateral tubal occlusion
     * Vasectomy - a vasectomy is highly effective contraception method provided the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used.
     * Male is sterile due to a bilateral orchiectomy.
     * Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual activity during the entire period of risk associated with the study drug. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient.

   List is not all inclusive. Prior to enrolment, the investigator is responsible for confirming patient will utilize highly effective forms of birth control in combination with a barrier method according to locally accepted standards during the protocol defined period.
   * agree not to breastfeed starting at screening and throughout the study period.
   * agree not to donate ova starting at screening and throughout the study period, and for 6 months after the final study drug administration.
10. Men must use a latex condom during any sexual contact with women of childbearing potential (WOCBP), even if they have undergone a successful vasectomy and must agree to avoid to father a child (while on therapy and for 6 months after the final study drug administration). In addition, their female partners of childbearing potential must use a highly effective method of birth control.
11. Male patient must not donate sperm starting at screening and throughout the study period and for 6 months after the final study drug administration.
12. Able to understand and willing to sign an informed consent form (ICF).
13. Institutional Review Board/Independent Ethics Committee-approved written informed consent as per national regulations must be obtained from the patient prior to any study-related procedures (including consent for withdrawal of prohibited medication, if applicable).

Exclusion Criteria:

Subject has previously been treated for AML; a treatment period with hydroxyurea to control WBC counts is allowed; prior treatment with a hypomethylating agent for MDS-EB is not allowed; prior treatment with erythropoiesis-stimulating agents or luspatercept for MDS is allowed.

2. Acute promyelocytic leukemia (APL) with t(15;17)(q24.1;q21.2); PML-RARA; or one of the other pathognomonic variant chromosomal translocations / fusion genes. 3. AML with BCR-ABL1; or myeloid blast crisis of CML. 4. Significant active cardiac disease within 3 months prior to the start of study treatment, including:

* New York Heart Association (NYHA) class III or IV congestive heart failure
* Myocardial infarction
* Unstable angina
* Severe cardiac arrhythmias
* Congenital long QT syndrome of family member with this condition QTcF >450 msec on screening electrogram for males and >470msec on screening electrogram for females (mean of triplicate recordings; calculated using Fridericia's correction). 5. Severe obstructive or restrictive ventilation disorder. 6. History of stroke or intracranial hemorrhage within 6 months prior to randomization.

  7. Clinical symptoms suggestive of active central nervous system (CNS) leukemia or known CNS leukemia. Evaluation of cerebrospinal fluid (CSF) during screening is only required if there is a clinical suspicion of CNS involvement by leukemia during screening. 8. Active infection, including hepatitis B or hepatitis C or Human Immunodeficiency Virus (HIV) infection, that is uncontrolled prior to first dose of study treatment and may interfere with the study objectives or which could expose the patient to undue risk through the participation in the clinical trial; an infection controlled with an approved antibiotic/ antiviral/ antifungal treatment that is not a strong or moderate CYP3A inducer is allowed. Patients with COVID-19 infection can be enrolled, if the patient has no symptoms and was tested negative twice by PCR test prior to inclusion in the trial. 9. Immediate life-threatening, severe complications of leukemia such as uncontrolled bleeding and/or disseminated intravascular coagulation. 10. Conditions that limit the ingestion or gastrointestinal absorption of orally administered drugs.

  11. Patient with a currently active second malignancy. Patients are not considered to have a currently active malignancy, if they have completed therapy and are considered by their physician to be at < 30% risk of relapse within one year. However, patients with the following history/concurrent conditions are allowed:
* Basal or squamous cell carcinoma of the skin;
* Carcinoma in situ of the cervix;
* Carcinoma in situ of the breast;
* Incidental histologic finding of prostate cancer. 12. Receipt of live, attenuated vaccine within 30 days prior to the study inclusion (NOTE: patient, if enrolled, should not receive live vaccine during the study and until 6 months after the therapy).

  13. Severe neurological or psychiatric disorder interfering with ability to give an informed consent.

  14. Known or suspected hypersensitivity to any of the anti-leukemic agents used.

  15. Participation in other prospective studies with anti-leukemic and/or investigational agents.

  16. Patient taking Dabigatran unless they can be transferred to other medications within ≥5 half-lives prior to dosing. Patients taking other P-gP transporter-sensitive medications (see Appendix H) should be properly monitored during the study if they cannot be transferred to other medications.

  17. Patient taking known strong cytochrome P450 (CYP) 3A4 inducers , unless they can be transferred to other medications within ≥5 half-lives prior to dosing. The patient is a pregnant or lactating woman, or plans to become pregnant during the study.

  19. Patient who has once been screened and randomized into this HO177 trial but was considered ineligible cannot re-enter this trial at a later date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2029-12-13 (Estimated); Study Completion 2031-07-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) in adult patients with newly diagnosed NPM1-mutated AML ineligible for intensive chemotherapy. | 58 months after last patient inclusion
  To assess if treatment with revumenib, in combination with azacitidine and venetoclax, prolongs overall survival (OS) measured from the date of randomization to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.

SECONDARY OUTCOMES:
Event-free survival (EFS) in adult patients with newly diagnosed NPM1-mutated AML ineligible for intensive chemotherapy. | 58 months after the first NPM1-mutated AML patient has been randomized
  Assess if treatment with revumenib, in combination with azacitidine and venetoclax, prolongs event-free survival (EFS); measured from the date of randomization to the date of treatment failure, hematologic relapse from CR/CRh or death from any cause, whichever occurs first. Treatment failure is defined as lack of obtaining either CR or CRh by week 24.
Rate of CR/CRh in adult patients with newly diagnosed NPM1mutated AML ineligible for intensive chemotherapy, | 58 months after the first randomized NPM1-mutated AML patient
  Defined as the proportion of NPM1-mutated AML patients who achieve CR or CRh at any time-point during protocol therapy.
Rate of CR in adult patients with newly diagnosed NPM1-mutated AML ineligible for intensive chemotherapy | 58 months after the first randomized NPM1-mutated AML patient
  Defined as the proportion of NPM1-mutated AML patients who achieve CR at any time-point during protocol therapy.
Rate of response (CRh and CR/CRi) in adult patients with newly diagnosed NPM1-mutated AML ineligible for intensive chemotherapy | 58 months after the first randomized NPM1-mutated AML patient
  Rate of response (CRh and CR/CRi) is defined as the proportion of patients with response at any time-point during protocol therapy.
Rates of CR, CR/CRh and CR/CRi without measurable residual disease (CRMRD-, CR/CRhMRD- and CR/CRiMRD-) | 58 months after the first randomized NPM1-mutated AML patient
  defined as the proportion of NPM1-mutated AML patients who achieve CR, CR/CRh and CR/CRi, respectively, and have no detectable MRD by molecular PCR at any time-point during protocol therapy
Time to achievement of response (CR, CR/CRh and CR/CRi) in adult patients with newly diagnosed NPM1-mutated AML ineligible for intensive chemotherapy ineligible for intensive chemotherapy | 58 months after the first randomized NPM1-mutated AML patient
  Defined as time from the date of randomization to until the 1st occurrence of response,
Duration of response (CR, CR/CRh and CR/CRi; DoR) in adult patients with newly diagnosed NPM1-mutated AML ineligible for intensive chemotherapy | 58 months after the first randomized NPM1-mutated AML patient
  Defined from the date of achievement of response until the date of hematologic relapse or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Gerwin Huls, MD, Principal Investigator — UMCG/ HOVON
Locations (67):
- Germany (29):
  - DE-Berlin-CAMPUSBENFRANKLIN, Berlin
  - DE-Berlin-CAMPUSVIRCHOW, Berlin
  - DE-Berlin-VIVANTESNEUKOLLN, Berlin
  - DE-Bochum-RUB, Bochum
  - DE-Bonn-UNIBONN, Bonn
  - DE-Braunschweig-KLINIKUMBRAUNSCHWEIG, Braunschweig
  - DE-Bremen-KBM, Bremen
  - DE-Darmstadt-KLINIKUMDARMSTADT, Darmstadt
  - DE-Essen-KEM, Essen
  - DE-Flensburg-MALTESER, Flensburg
  - DE-Frankfurt-KLINIKUMFRANKFURT, Frankfurt
  - DE-Freiburg-UNIKLINIKFREIBURG, Freiburg im Breisgau
  - DE-Greifswald-UNIGREIFSWALD, Greifswald
  - DE-Hamburg-ASKLEPIOSSTGEORG, Hamburg
  - DE-Hamburg-UKE, Hamburg
  - DE-Hannover-MHHANNOVER, Hanover
  - DE-Hannover-SILOAHKRH, Hanover
  - DE-Heilbronn-SLK General Information, Heilbronn
  - DE-Herne-MARIENHOSPITALHERNE, Herne
  - DE-Karlsruhe-KLINIKUMKARLSRUHE, Karlsruhe
  - DE-Mainz-UNIMEDIZINMAINZ, Mainz
  - DE-Minden-MUEHLENKREISKLINKEN, Minden
  - DE-München-IRZTUM, München
  - DE-Oldenburg-KLINIKUMOLDENBURG, Oldenburg
  - DE-Potsdam-BERGMANN, Potsdam
  - DE-Stuttgart-KLINIKUMSTUTTGART, Stuttgart
  - DE-Tübingen-MEDUNITUEBINGEN, Tübingen
  - DE-Ulm-UNIKLINKULM, Ulm
  - DE-Wuppertal-HELIOSGESUNDHEIT, Wuppertal
- Netherlands (20):
  - NL-Den Bosch-JBZ, 's-Hertogenbosch
  - NL-Amersfoort-MEANDERMC, Amersfoort
  - NL-Amsterdam-OLVG, Amsterdam
  - NL-Amsterdam-VUMC, Amsterdam
  - NL-Arnhem-RIJNSTATE, Arnhem
  - NL-Breda-AMPHIA, Breda
  - NL-Delft-RDGG, Delft
  - NL-Eindhoven-MAXIMAMC, Eindhoven
  - NL-Enschede-MST, Enschede
  - NL-Goes-ADRZ, Goes
  - NL-Groningen-UMCG, Groningen
  - NL-Leeuwarden-MCL, Leeuwarden
  - NL-Leiden-LUMC, Leiden
  - NL-Maastricht-MUMC, Maastricht
  - NL-Nieuwegein-ANTONIUS, Nieuwegein
  - NL-Nijmegen-RADBOUDUMC, Nijmegen
  - NL-Rotterdam-ERASMUSMC, Rotterdam
  - NL-Den Haag-HAGA, The Hague
  - NL-Utrecht-UMCUTRECHT, Utrecht
  - NL-Zwolle-ISALA, Zwolle
- United Kingdom (18):
  - Belfasttrust, Belfast
  - Birmingham-QE, Birmingham
  - Blackpool Victoria, Blackpool
  - UH Bristol, Bristol
  - University Hospital of Wales, Cardiff
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St. James UH, Leeds
  - University Hospitals of Leicester NHS Trust, Leicester
  - University of Liverpool, Liverpool
  - King's College Hospital, London
  - St Bartholomew's Hospital, London
  - Christie NHS Foundation Trust, Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Churchill Hospital, Oxford, Oxford
  - Southampton General Hospital, Southampton
  - The Royal Marsden NHSFT, Sutton
  - New cross hospital wolverhampton, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
According to the current publication policy the protocol and Statistical Analysis Plan ( SAP) will be shared. The principal Investigators can be contacted for IPD sharing after the publication of the study results. According to 'HOVON sample and/or Data request Form' the HOVON director; chair of the HOVON Acute Myeloid Leukemic working group, the study PI and Coordinating Investigator should approve data/sample sharing.
Supporting Information: Study Protocol, SAP
Time Frame: After the publication of primary endpoint analysis

REFERENCES:
- See also: HOVON website — http://hovon.org